CLINICAL TRIAL: NCT01266252
Title: Dexmedetomidine Pharmacokinetics - Pharmacodynamics in Mechanically Ventilated Neonates With Single-organ Respiratory Failure (NEODEX).
Brief Title: Dexmedetomidine in Mechanically Ventilated Neonates With Single-Organ Respiratory Failure.
Acronym: NEODEX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC/2010/786
Record Dates: First submitted 2010-12-22; First posted 2010-12-24 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Mechanically-ventilated Neonates With Single-organ Respiratory Failure
Keywords: neonates; single organ respiratory failure
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dexmedetomidine (Experimental)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine will be given maximal 72 hours. In case analgosedation is still needed after stop of the dexmedetomidine infusion, the treatment is switched to conventional analgosedation regimens.
  Additional drugs are given to every inadequately sedated-painful patient (assessed by regular Comfort-neo and Numeric Rating Scale scoring). In case of oversedation or adverse drug events (hypotension, bradycardia), a downtitration (or stop) of the dexmedetomidine infusion is needed.

SUMMARY:
Clinical experience with dexmedetomidine in the paediatric population is limited. Critical illness can affect drug pharmacokinetics and -dynamics; the investigators cannot simply extrapolate adult data for use in children but the investigators are in need of data on pharmacokinetics and pharmacodynamics in every paediatric subpopulation.

DETAILED DESCRIPTION:
Currently, dexmedetomidine is approved by the United States Food and Drug Administration (FDA) for short-term analgosedation (<24h) in mechanically-ventilated critical care adult patients and sedation of non-intubated adult patients prior to and/or during surgical and other procedures. Trials are underway to investigate its pharmacokinetics, clinical efficacy and safety in long-term use. Clinical experience with dexmedetomidine in the paediatric population is limited. Moreover, during childhood many developmental changes take place with consequences on drug exposure and drug response. Finally, critical illness itself can affect drug pharmacokinetics and -dynamics. Therefore, the investigators cannot simply extrapolate adult data for use in children but the investigators are in need of data on pharmacokinetics and pharmacodynamics in every paediatric subpopulation.

ELIGIBILITY:
Inclusion Criteria:

* patient age less than 1 month (Male/Female) (step-down strategy for age)

  * first included patients (n=30): postmenstrual age >= 34 weeks (near-term neonates)
  * following included patients (n=30) : postmenstrual age >= 25 weeks and < 34 weeks (preterm neonates)
* patients with single-organ respiratory failure in need for analgosedation (guidance : Comfort neo score >14 or Numeric Rating Scale (NRS) score Pain (P)/Comfort (C)>4)
* patients admitted to the neonatal intensive care unit
* expected to require at least 20 hours of mechanical ventilation

Exclusion Criteria:

* patients with neurologic conditions that prohibit an evaluation of adequate analgosedation
* no arterial catheter in place at inclusion
* patients who have received another investigational drug within 30 days
* patients on continuous infusion with neuromuscular blockers
* patients with a life expectancy <72 hours
* patients with a known allergy to fentanyl
* congenital or acquired heart block (grade 3)
* sustained bradycardia
* haemodynamically unstable patients (definition : Mean Arterial Pressure (MAP) lower than : postmenstrual age (in weeks) - 5 millimeter Hg, eventually under dopamine infusion max. 16 mcg/kilogram/minute and/or dobutamine infusion maximal 16 mcg/kilogram/minute)
* patients with significant renal insufficiency (creatinine plasma level >1.5 milligram/deciliter)
* patients with significant hepatic insufficiency (as estimated by local investigators)
* previous treatment with α2-adrenoreceptor agonist clonidine within 14 days
* absence of parental consent

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2011-07-28 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2018-04-10 (Actual)

PRIMARY OUTCOMES:
pharmacokinetic parameters | 72 hours
  Pharmacokinetic parameters of dexmedetomidine infusion in mechanically ventilated neonates with single-organ respiratory failure.
Covariates | 72 hours
  Covariates contributing to a variability in exposure and response to dexmedetomidine.

SECONDARY OUTCOMES:
level of analgosedation | 72 hours
  Preliminary knowledge on the level of analgosedation provided by dexmedetomidine.
safety issues | 72 hours
  Preliminary knowledge of safety issues concerning systolic and diastolic blood pressure, heart rate, respiratory rate, oxygen saturation, temperature are assessed baseline and at least per hour reassessed after starting the dexmedetomidine infusion.
variability due to the Cytochrome P450 2A6 (CYP2A6) and Uridine diphosphate (UDP)-glucuronosyltransferase genotype | 72 hours
  Knowledge of the contribution of the Cytochrome P450 2A6 (CYP2A6) and Uridine diphosphate (UDP)-glucuronosyltransferase genotype (covariate) to the variability in exposure and response to dexmedetomidine.

CONTACTS AND LOCATIONS:
Overall Officials: Koenraad Smets, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (3):
- Belgium (3):
  - AZ Bruges, Bruges
  - Ghent University Hospital, Ghent
  - UZ Leuven, Leuven

REFERENCES:
- See also: Related Info — http://www.uzgent.be